CLINICAL TRIAL: NCT01493076
Title: Safety and Efficacy of a New Baby-sphincterotome for Cannulation and Pre-cut in Failed Selective Wire-guided Bile Duct Access
Brief Title: Safety and Efficacy of a Newly Developed Baby-sphincterotome for Bile Duct Cannulation
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Andrea Riphaus, Assistant medical director, Ruhr University of Bochum
Other Study IDs: Baby-S 2011
Record Dates: First submitted 2011-11-20; First posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Bile Duct Diseases
Keywords: ERCP; Cannulation; Precut; Mini-spincterotome
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Baby-S group: The baby-sphincterotome was in patients in whom biliary sphincterotomy was clinically indicated but in whom after standard techniques to gain biliary access had failed (study population).
  Interventions: Device: Primary cannulation/precut sphincterotomie with the Baby-S

INTERVENTIONS:
Device: Primary cannulation/precut sphincterotomie with the Baby-S — At the papilla the ankle for cannulation was optimized due to changes of the position of the sphincterotome, its lay in the working channel and the tension of the "Albaran"-lever and the cutting wire. After successful cannulation, the catheter with the sphincterotome inside was slightly pushed into the duct. If necessary, the baby-sphincterotome was replaced with a guide wire and than conventional endoscopic sphincterotomie was completed with a standard traction-type sphincterotome.
  Other Names: Easy-Cut®, MTW, Wesel, Germany

SUMMARY:
Precut-sphincterotomy is a well established alternative after repeated futile attempts for common bile duct (CBD) cannulation with standard catheters and/or guide-wires fail. Commonly used devices instruments for pre-cutting are the needle-knife and the Erlangen-type precut-sphincterotome. In 1996 a so called "baby-sphincterotome" (Easy-Cut®, MTW, Wesel, Germany) with a pre-shaped-bended (to facilitate biliary access) small-calibre 3-French tip was developed, which enables cannulation and pre-cutting in one step. Here the investigators report on the clinical evaluation of this device.

DETAILED DESCRIPTION:
Interventional procedures at the bile or pancreatic duct require selective cannulation of the desired duct and sometimes endoscopic sphincterotomy (ES). If it is not possible to achieve selective access to the desired duct, which occurs in about 10-33 % of the cases (1-4), the next step to ensure selective cannulation is a so-called pre-cut procedure (5-8). For this approach a needle knife or an Erlangen-type sphincterotome are used to perform pre-cut sphincterotomy (PCS). This pre-cut technique has been shown to be effective especially to obtain selective bile duct access in the majority of the cases whenever standard cannulation techniques fail. However, the reported complication rate for PCS is substantially higher than for conventional ES (9), but may be outweighed by the clinical benefits. A limitation of the PCS-procedure is the need to use a dedicated instrument (either the needle knife or the Erlangen-type sphincterotome) for this indication. After completion of the pre-cut procedure routinely the attempt access to the desired duct has to be performed with other accessories since most pre-cut-sphincterotomes did do not allow contrast injection or guide-wire insertion. A change of instruments before and after PCS prolongs procedure time and increases cost. Therefore a "universal" instrument designed for both bile duct cannulation and precutting would substantially simplify the procedure.

In 1999 the investigators described a newly developed "baby"-sphincterotome that combines the features of a cannulating catheter and Erlangen-type precut-papillotome. In a first series of patients this device was found to be useful for direct cannulation as well as for precut procedures (10).

The aim of this trial was to investigate the safety and efficacy of this newly developed baby-sphincterotome in cases of failed selective wire-guided bile duct cannulation in a large cohort of patients.

Inclusion criteria were: evidence for bile duct obstruction with a visible stone or tumor, dilated common bile duct > 7 mm (or > 9 mm in cholecystectomised patients) by ultrasonography and CT-scan or MRCP/EUS, an elevated serum bilirubin level > 1.4 mg/dl, and serum alkaline phosphatase > 200 U/l with clinical suspicion of obstruction without evidence for cholestatic liver disease.

Patients with severe coagulation disorders or distorted anatomy of the major papilla (malignant infiltration of the papilla, papillary porus not identifiable, impacted stone) and patients with former gastro-duodenal resection (e.g. BII-anatomy) were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Evidence for bile duct obstruction with a visible stone or tumor, dilated common bile duct > 7 mm (or > 9 mm in cholecystectomised patients) by ultrasonography and CT-scan or MRCP/EUS, an elevated serum bilirubin level > 1.4 mg/dl, and serum alkaline phosphatase > 200 U/l with clinical suspicion of obstruction without evidence for cholestatic liver disease.

Exclusion Criteria:

* Patients with severe coagulation disorders or distorted anatomy of the major papilla (malignant infiltration of the papilla, papillary porus not identifiable, impacted stone) and patients with former gastro-duodenal resection (e.g. BII-anatomy) were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Use of the baby-sphincterotome for cannulation and pre-cut in cases of failed selective wire-guided bile duct access.
Sampling Method: Probability Sample
Enrollment: 1886 (Actual)
Dates: Start 2000-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with successfull bile duct cannulation | Time-to-Event Outcome Measures from the beginning of the intervention until the end of the endoscopic procedure, participants will be followed for the duration of hospital stay, an expected average of 3-5 days
  The baby-sphincterotome was used in patients in whom biliary sphincterotomy was clinically indicated but in whomafter standard techniques to gain biliary access had failed (study population).

SECONDARY OUTCOMES:
Postinterventional compilation rate (bleeding, pancreatitis) | Immediate or delayed complications. Time-to-Event Outcome Measures: from the beginning of the intervention till signs bleeding or panceatitis will occur. Participants will be followed for the duration of hospital stay, an expected average of 3-5 days
  The severity of post-ERCP-pancreatitis was graded according to the Cotton criteria (Cotton et al.). Mild post-sphincterotomy bleeding was any bleeding episode detected after ES or PCS that necessitatinge an endoscopic maneuver like injection or clipping whithin the same session.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Riphaus, MD, PhD, Principal Investigator — Ruhr University Bochum, Department of Medicine; Riphaus Andrea, MD, PhD, Principal Investigator — Department of Medicine, Ruhr University Bochum

REFERENCES:
- [Background] Foutch PG. A prospective assessment of results for needle-knife papillotomy and standard endoscopic sphincterotomy. Gastrointest Endosc. 1995 Jan;41(1):25-32. doi: 10.1016/s0016-5107(95)70272-5. PMID 7698621
- [Background] Seifert H, Binmoeller KF, Schmitt T, Dietrich CF, Zipf A, Caspary WF, Wehrmann T. [A new papillotome for cannulation, pre-cut or conventional papillotomy]. Z Gastroenterol. 1999 Dec;37(12):1151-5. German. PMID 10666838